CLINICAL TRIAL: NCT01321853
Title: Home Care Medication Management Program for the Frail Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Wisconsin, Milwaukee (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 144PG09; 5R01NR008911 (NIH)
Record Dates: First submitted 2011-03-15; First posted 2011-03-24 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Illness; Cognitive Impairment
Keywords: Home health care; Medication Management; Cognitive impairment; Medication adherence; Older adults; Care Coordination management
MeSH Terms: conditions — Chronic Disease; Cognitive Dysfunction; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Machine and NCC (Experimental): Medications dispensed to subject via MD2 machine and nurse care coordination used to coordinate care among providers and fill machine at least every 2 weeks.
  Interventions: Other: MD2 machine and nurse care coordination
- Medplanner and NCC (Experimental): Medications loaded in medplanner by nurse care coordinator who coordinates care among providers and visits subject at least every 2 weeks
  Interventions: Other: Medplanner and Nurse Care Coordination
- Usual Care Group (No Intervention): Admitted post home health care with no intervention.

INTERVENTIONS:
Other: MD2 machine and nurse care coordination — MD2 machine filled at least every 2 weeks and subjects monitored for changes in condition. Additional visits made as needed. Care is coordinated with other providers such as the primary care physician and pharmacist.
  Arms: Machine and NCC
Other: Medplanner and Nurse Care Coordination — Medications are dispensed via a medplanner filled by a nurse at least every 2 weeks and subjects monitored for changes in condition. Additional visits made as needed. Care is coordinated with other providers such as the primary care physician and pharmacist.
  Arms: Medplanner and NCC

SUMMARY:
The purpose of this study is to determine whether a home care medication management program which includes nurse coordination and use of the MD.2 medication-dispensing machine will affect older adults' health outcomes, satisfaction, use of health care services, and health care costs over a one year period. The investigators propose a longitudinal three group repeated measures design, enrolling, and randomly assigning, clients who are discharged from a home health care agency with documented problems in medication management. One group will receive the MD.2 medication dispensing device and nurse coordination, the second group will receive a Medplanner: a simple box that has separate compartments for individual medication times over the course of a week plus nurse coordination, and the final group will receive Usual Care.

The study hypotheses are the following:

H1: With respect to health status outcomes, the MD.2 group will exhibit a more positive trajectory in physical and mental health status, functional status, cognitive status and depressive symptoms over the course of a year than will the Medplanner Group.

H2: With respect to health status outcomes, the Medplanner Group will exhibit a more positive trajectory in physical and mental health status, functional status, cognitive status and depressive symptoms over the course of a year than will the Usual Care Group.

H3: The rate of hospitalization, hospital days and emergency department visits will be significantly lower for the MD.2 Group as compared to the Medplanner Group.

H4: The rate of hospitalization, hospital days and emergency department visits will be significantly lower for the Medplanner Group as compared to the Usual Care Group.

H5: The nursing home admission rate will be significantly lower for the MD.2 Group as compared to the Medplanner Group.

H6: The nursing home admission rate will be significantly lower for the Medplanner Group as compared to the Usual Care Group.

H7: The total cost of care will be significantly lower for the MD.2 Group as compared to the Medplanner Group.

H8: The total cost of care will be significantly lower for the Medplanner Group as compared to The Usual Care Group.

H9: There will be incremental savings in terms of costs per quality adjusted life year (QALY) gained in the MD.2 group compared with the Medplanner Group.

H10: There will be incremental savings in terms of costs per QALY gained in the Medplanner group compared with the Usual Care Group.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Medicare Primary Payer
* Impaired Medication Management ability as indicated by a score of 1 or higher on OASIS discharge assessment item M0780
* Impaired Cognitive Functioning but able to follow directions with prompting as indicated by a score of 1 or 2 on OASIS discharge assessment item M0560
* working telephone line
* Discharge from home health care

Exclusion Criteria:

* Not English speaking
* Terminal diagnosis or hospice care
* Use of other device for medications
* Medicare via managed care
* Use of private home care agency for medication management

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Geriatric Depression Scale | 12 months
  The Geriatric Depression Scale (GDS) was developed to identify depression in older adults. The original GDS was 30 questions, however, fifteen- and five-question versions also exist. When tested on the oldest old in the community, the 15-item scale was demonstrated to have favorable reliability and validity results. Impaired cognitive function (MMSE < 28) reduced the tool's specificity, but sensitivity was not affected by lower MMSE scores. The tool is scored into depression categories of "none/mild", "moderate" and "major".
Physical Performance Test (PPT) | 12 months
  This functional status test has demonstrated reliability and validity, is easy to administer, can be performed in a reasonable period of time, and imposes little burden on the individual being tested. Even men and women with mild to moderate dementia are capable of understanding the test and performing activities reliably. There are 7 items on the test that range in difficulty from very easy to perform (writing a sentence) to challenging (picking up a penny), thus encompassing a spectrum of physical capabilities.
SF-36 Health Survey | 12 months
  This tool is a widely used generic health status questionnaire measuring eight dimensions of health status: physical functioning, role limitations due to physical health problems, bodily pain, social functioning, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. In addition, the SF-36 can be transformed into a Health State Utility Index that allows for health improvements to be stated in terms of quality adjusted life years (QALYs) gained.
Mental Mental Status Exam (MMSE) | 12 months
  This 11-item measure screens for cognitive abilities in the domains of orientation, memory, attention, recall, language and visual/spatial orientation. The MMSE may be a categorical or continuous-level variable. When used as a categorical variable, the MMSE is broken down into 4 levels: (a) score range 24-30 is considered within normal limits (WNL), (b) score range of 18-23 is considered mild cognitive impairment, (c) score range of 12-17 is considered moderate cognitive impairment, and (d) a score range of 11 or less is considered to be severe cognitive impairment.
Hospitalization | 12 month enrollment period
  Medicare claims data will be the source of information for this measure.
Hospital Days | 12 Month Enrollment Period
  Medicare claims data will be the source of information for this measure.
Emergency Department Visits | 12 month Enrollment Period
  Medicare claims data will be the source of information for this measure.
Medicare Costs | 12 Month Enrollment Period
  Medicare claims data will be the source of information for this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Marek, PhD, Principal Investigator — Arizona State University
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Marek KD, Stetzer F, Ryan PA, Bub LD, Adams SJ, Schlidt A, Lancaster R, O'Brien AM. Nurse care coordination and technology effects on health status of frail older adults via enhanced self-management of medication: randomized clinical trial to test efficacy. Nurs Res. 2013 Jul-Aug;62(4):269-78. doi: 10.1097/NNR.0b013e318298aa55. PMID 23817284